CLINICAL TRIAL: NCT04404946
Title: Colloid Co-hydration and Vasoconstrictor Infusion for Prevention of Postspinal Hypotension During Elective Cesarean Section. A Comparative Study
Brief Title: Colloid Co-hydration and Vasoconstrictor Infusion for Prevention of Hypotension During Cesarean Section
Acronym: annie-zoe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aretaieion University Hospital (Other)
Responsible Party: Principal Investigator, Dr Kassiani Theodoraki, Professor of Anesthesiology, Aretaieion University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 196/25-02-2020
Record Dates: First submitted 2020-05-22; First posted 2020-05-28 (Actual); Last update posted 2021-06-15 (Actual); Status verified 2021-06

CONDITIONS: Hypotension Symptomatic; Vasoconstriction; Cesarean Section Complications; Obstetric Anesthesia Problems

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- phenylephrine infusion (Active Comparator): fixed-rate phenylephrine infusion
  Interventions: Other: phenylephrine infusion
- norepinephrine infusion (Active Comparator): fixed-rate norepinephrine infusion
  Interventions: Other: norepinephrine infusion
- placebo infusion (Placebo Comparator): normal saline infusion
  Interventions: Other: placebo infusion

INTERVENTIONS:
Other: phenylephrine infusion — in parturients allocated to the phenylephrine group, a phenylephrine infusion will be started as soon as spinal anesthesia is initiated
  Other Names: medication used for blood pressure maintenance
  Arms: phenylephrine infusion
Other: norepinephrine infusion — in parturients allocated to the norepinephrine group, a norepinephrine infusion will be started as soon as spinal anesthesia is initiated
  Other Names: medication used for blood pressure maintenance
  Arms: norepinephrine infusion
Other: placebo infusion — in parturients allocated to the placebo group, a normal saline infusion will be started as soon as spinal anesthesia is initiated
  Other Names: medication used for blood pressure maintenance
  Arms: placebo infusion

SUMMARY:
This will be a double-blind randomized study, aiming at investigating a fixed rate phenylephrine infusion versus a fixed rate norepinephrine infusion versus placebo in combination with co-hydration with colloids for the prevention of maternal hypotension in elective cesarean section

DETAILED DESCRIPTION:
Neuraxial techniques are the anesthetic techniques of choice in contemporary obstetric anesthesia practice, with a definitive superiority as compared to general anesthesia, since, by their use, serious complications involving the airway can be avoided.Spinal anesthesia has become the favorable technique for both elective and emergency cesarean section due to a quick and predictable onset of action, however, it can be frequently complicated by hypotension, with incidence exceeding 80% occasionally.

The aim of the current randomized controlled double-blinded trial was to compare the effect of a fixed-rate norepinephrine infusion versus a fixed-rate phenylephrine infusion versus placebo in parturients subjected to elective cesarean section under combined spinal-epidural anesthesia. All parturients will also receive colloid co-hydration.

ELIGIBILITY:
Inclusion Criteria:

* adult parturients, American Society of Anesthesiologists (ASA) I-II,
* singleton gestation>37 weeks
* elective cesarean section

Exclusion Criteria:

* Body Mass Index (BMI) >40 kg/m2
* Body weight <50 kg
* Body weight>100 kg
* height<150 cm
* height>180 cm
* multiple gestation
* fetal abnormality
* fetal distress
* active labor
* cardiac disease
* pregnancy-induced hypertension
* thrombocytopenia
* coagulation abnormalities
* use of antihypertensive medication during pregnancy
* communication or language barriers
* lack of informed consent
* contraindication for regional anesthesia

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 120 (Actual)
Dates: Start 2020-05-23 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
incidence of bradycardia | intraoperative
  any incidence of maternal bradycardia (heart rate<60/min) will be recorded
incidence of hypotension | intraoperative
  any occurence of hypotension (systolic blood pressure<80% of baseline) throughout the operation will be recorded

SECONDARY OUTCOMES:
need for vasoconstrictor | intraoperative
  any need for vasoconstrictor during the operation will be recorded
type of vasoconstrictor administered | intraoperative
  phenylephrine versus ephedrine
number of bolus doses of vasoconstrictor administered | intraoperative
  number of interventions to maintain systolic blood pressure within the set limits will be recorded
total dose of vasoconstrictor administered | intraoperative
  total dose in mg for ephedrine or μg for phenylephrine administered
incidence of hypertension | intraoperative
  any incidence of systolic blood pressure>120% of baseline will be recorded
need for atropine | intraoperative
  any need for atropine during the operation because of bradycardia will be recorded
modification or cessation of the infusion | intraoperative
  any requirement for modification or cessation of the infusion due to reactive hypertension or bradycardia will be recorded
incidence of nausea/vomiting | intraoperative
  any occurence of nausea and/or vomiting during the operation will be recorded
Neonatal Apgar score at 1 minutes | 1 minute post delivery
  Neonatal Apgar score will be recorded at 1 minutes after delivery. The Apgar score is determined by evaluating the newborn baby on five simple criteria on a scale from zero to two, then summing up the five values thus obtained. The resulting Apgar score ranges from zero to 10. Scores 7 and above are generally normal; 4 to 6, fairly low; and 3 and below are generally regarded as critically low and cause for immediate resuscitative efforts.
Neonatal Apgar score at 5 minutes | 5 minutes post delivery
  Neonatal Apgar score will be recorded at 5 minutes after delivery. The Apgar score is determined by evaluating the newborn baby on five simple criteria on a scale from zero to two, then summing up the five values thus obtained. The resulting Apgar score ranges from zero to 10. Scores 7 and above are generally normal; 4 to 6, fairly low; and 3 and below are generally regarded as critically low and cause for immediate resuscitative efforts.
neonatal blood gases | 1 minute post delivery
  fetal cord blood analysis will be performed immediately post-delivery
glucose in neonatal blood | 1 minute post delivery
  glucose will be measured in the cord blood gas sample taken immediately post-delivery
adrenaline in neonatal blood | 5 minutes post delivery
  an amount of the umbilical artery cord blood sampled from every neonate will be sent for lab measurements
noradrenaline in neonatal blood | 5 minutes post delivery
  an amount of the umbilical artery cord blood sampled from every neonate will be sent for lab measurements

OTHER OUTCOMES:
cardiac output | intraoperative
  cardiac output via non-invasive device (Nexfin) will be measured intraoperatively
stroke volume | intraoperative
  stroke volume via non-invasive device (Nexfin) will be measured intraoperatively
systemic vascular resistance | intraoperative
  systemic vascular resistance via non-invasive device (Nexfin) will be measured intraoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Kassiani Theodoraki, PhD, DESA, Principal Investigator — Aretaieion University Hospital
Locations (1):
- Aretaieion University Hospital, Athens, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Langesaeter E, Dyer RA. Maternal haemodynamic changes during spinal anaesthesia for caesarean section. Curr Opin Anaesthesiol. 2011 Jun;24(3):242-8. doi: 10.1097/ACO.0b013e32834588c5. PMID 21415724
- [Background] Ngan Kee WD. Prevention of maternal hypotension after regional anaesthesia for caesarean section. Curr Opin Anaesthesiol. 2010 Jun;23(3):304-9. doi: 10.1097/ACO.0b013e328337ffc6. PMID 20173633
- [Background] Kinsella SM, Carvalho B, Dyer RA, Fernando R, McDonnell N, Mercier FJ, Palanisamy A, Sia ATH, Van de Velde M, Vercueil A; Consensus Statement Collaborators. International consensus statement on the management of hypotension with vasopressors during caesarean section under spinal anaesthesia. Anaesthesia. 2018 Jan;73(1):71-92. doi: 10.1111/anae.14080. Epub 2017 Nov 1. No abstract available. PMID 29090733
- [Background] Mets B. Should Norepinephrine, Rather than Phenylephrine, Be Considered the Primary Vasopressor in Anesthetic Practice? Anesth Analg. 2016 May;122(5):1707-14. doi: 10.1213/ANE.0000000000001239. No abstract available. PMID 27101504
- [Background] Carvalho B, Dyer RA. Norepinephrine for Spinal Hypotension during Cesarean Delivery: Another Paradigm Shift? Anesthesiology. 2015 Apr;122(4):728-30. doi: 10.1097/ALN.0000000000000602. No abstract available. PMID 25654435
- [Background] Sen I, Hirachan R, Bhardwaj N, Jain K, Suri V, Kumar P. Colloid cohydration and variable rate phenylephrine infusion effectively prevents postspinal hypotension in elective Cesarean deliveries. J Anaesthesiol Clin Pharmacol. 2013 Jul;29(3):348-55. doi: 10.4103/0970-9185.117106. PMID 24106360
- [Background] Gunusen I, Karaman S, Ertugrul V, Firat V. Effects of fluid preload (crystalloid or colloid) compared with crystalloid co-load plus ephedrine infusion on hypotension and neonatal outcome during spinal anaesthesia for caesarean delivery. Anaesth Intensive Care. 2010 Jul;38(4):647-53. doi: 10.1177/0310057X1003800337. PMID 20715726
- [Background] Kulkarni KR, Naik AG, Deshpande SG. Evaluation of antihypotensive techniques for cesarean section under spinal anesthesia: Rapid crystalloid hydration versus intravenous ephedrine. Anesth Essays Res. 2016 Sep-Dec;10(3):637-642. doi: 10.4103/0259-1162.191118. PMID 27746565